CLINICAL TRIAL: NCT01865435
Title: IN UTERO SMOKING AND PREMATURE CELLULAR SENESCENCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2012-A01655-38; 2012-52 (Other: AP HM)
Record Dates: First submitted 2013-05-27; First posted 2013-05-30 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- new borns (Experimental)
  Interventions: Genetic: cord blood sample

INTERVENTIONS:
Genetic: cord blood sample

SUMMARY:
Actually, there is an increasing number of arguments for a premature origin of chronic adult's diseases, as the chronic obstructive pulmonary disease (COPD). Several factors interacting with the foetal or postnatal lung growth are associated with early and long-lasting respiratory functional changes susceptible to contribute very significantly to the arisen of a COPD in the adulthood. It is possible that these situations reflect phenomena of premature cellular senescence, recently involved in the physiopathology of the COPD. An in utero exposition to cigarette smoking is one of these situations, because it is known to induce, not only functional respiratory changes, but also multiple diseases in the child which could testify of cellular ageing phenomena.

Our project aims to demonstrate that in utero smoking is associated with markers of premature cellular senescence in newborn children

The study will be driven in human newborn child's, with comparison of the length of the telomeres in circulating lymphocytes (umbilical blood is collected), according to the exposure in in utero smoking and also according to the degree of hypotrophy. This study will be a pilot study completed by an animal experimental study.

ELIGIBILITY:
Inclusion Criteria:

* Born weight upper or equal to the 10th percentile and absence of smoking declared by the mother
* Born weight lower than the 10th percentile and absence of smoking declared by the mother
* Born weight upper or equal to the 10th percentile and smoking declared by the mother of at least 5 cigarettes a day
* Born weight lower than the 10th percentile and smoking declared by the mother of at least 5 cigarettes a day

Exclusion Criteria:

* Gestationnel age 37 LIMITED COMPANIES
* Low(Weak) declaratory(declarative) maternal smoking (1 in 4 cigarettes a day)
* Pathologies associated by the newborn child (deformations, foetal suffering, infection maternofœtale, respiratory distress syndrome)

Max Age: 27 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2014-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
cord blood samples | 12months

CONTACTS AND LOCATIONS:
Overall Officials: LOIC MONDOLONI, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France